CLINICAL TRIAL: NCT01551407
Title: Open Prospective Within Patient, Phase IIa Study of Hexvix Flexible Cystoscopy and White Light Cystoscopy in the Detection of Bladder Cancer After 30 Minutes Instillation of Hexvix in Patients With Known or Suspicion of Bladder Cancer
Brief Title: Detection of Bladder Tumors After 30 Min Instillation of Hexvix
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow inclusion rate
Sponsor: Photocure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PC B202/11
Record Dates: First submitted 2012-03-02; First posted 2012-03-12 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Bladder Cancer
Keywords: Hexvix; bladder cancer; cystoscopy; Patients with known or suspicion of bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Hexvix — 50 ml Hexvix liquid instilled once into the bladder for 30 minutes prior to cystoscopy

SUMMARY:
The objective of the study is to compare Hexvix® flexible cystoscopy and white light flexible cystoscopy in the detection of histological confirmed bladder tumor lesions defined as dysplasia; CIS; Ta; T1; and ≥ T2 after 30 minutes intravesical instillation of Hexvix®.

DETAILED DESCRIPTION:
This study is an open, prospective, within patient, controlled, multi-center, Phase IIa study in patients with bladder cancer.

The bladder of all patients will be instilled with 50 mL Hexvix® 8 mM solution and evacuated after 30 minutes. After bladder evacuation, the bladder will be examined under white light cystoscopy using the Karl Storz flexible videocystoscope. Tumors visible under white light will be mapped. Then the bladder is evaluated with blue light and lesions seen by blue light will be mapped. Biopsies of all visible tumors will be taken using both white and blue light prior to resection of all lesions.

ELIGIBILITY:
Inclusion Criteria:

The patients should be indicated for a transurethral resection of the bladder (TURB) based on an outpatient cystoscopy and fulfil the following inclusion criteria:

* Patients with multiple bladder tumors, defined as ≥2 lesions, based on an outpatient cystoscopy.
* Patients with known urinary urge symptoms or patients who have problems or pain holding back the urine for a time longer than 30 minutes.
* Age 18 years or above

Exclusion Criteria:

* Patients with known tumors in the prostatic urethra or distal urethra
* Gross haematuria. (Note: Gross haematuria is defined as a heavy bladder bleed resulting in marked amounts of blood in the urine, which may interfere with fluorescence cystoscopy. Where the bleed is light, the patient should not be excluded if in the investigator's opinion, rinsing during cystoscopy will alleviate the possible interference with fluorescence cystoscopy).
* Patient with porphyria.
* Hypersensitivity to the active substance or to any of the excipients of the solvent
* Participation in other clinical studies with investigational drugs either concurrently or within the last 30 days.
* Women of child-bearing potential meaning that only post-menopausal women, women who had their ovaries removed, and women who are otherwise physically unable to bear children can be included.
* Patients who have received BCG or chemotherapy within three months prior to study inclusion.
* Conditions associated with a risk of poor protocol compliance.
* Patient is the investigator or any sub investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the clinical study.
* Patients unlikely to comply with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of lesions | An average of 15 min (during cystoscopy)

SECONDARY OUTCOMES:
Drug related adverse events | From time of drug instillation until 24 hours after cystoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Karl, MD, Principal Investigator — Department of Urology, LMU Munich, Germany
Locations (1):
- LMU Munich, Munich, Munich, Germany